CLINICAL TRIAL: NCT02790918
Title: Noninvasive Diagnosis of Pulmonary Hypertension Using Three-dimensional Interventricular Septal Curvedness From Cardiac Magnetic Resonance Images
Brief Title: Diagnosis of Pulmonary Hypertension Using Cardiac Magnetic Resonance Images
Status: Completed | Type: Observational
Sponsor: National Heart Centre Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2013/290/C
Record Dates: First submitted 2016-05-30; First posted 2016-06-06 (Estimated); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary Hypertension; MRI
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Diagnosed Pulmonary Hypertension: Patients will undergo the following studying procedures: Cardiovascular Magnetic Resonance Imaging (CMRI) and 6MWT.
  Interventions: Other: 6MWT; Other: Cardiovascular Magnetic Resonance Imaging (CMRI)
- Healthy Volunteer: Healthy Volunteer will undergo the following studying procedures: Cardiovascular Magnetic Resonance Imaging (CMRI) and 6MWT.
  Interventions: Other: 6MWT; Other: Cardiovascular Magnetic Resonance Imaging (CMRI)

INTERVENTIONS:
Other: 6MWT — Each patient will also receive 6MWT at cardiovascular rehabilitation and preventive cardiology laboratory. Besides the distance covered in meters or converted measure (such as feet) over 6 minutes, a portable metabolic system is used to measure oxygen uptake during exercise (VO2 testing) for each patient.
Other: Cardiovascular Magnetic Resonance Imaging (CMRI) — MRI uses interaction of the magnetic properties of body tissues with strong magnetic fields to create images; for about 1 hour. Several sets of images are needed. No injection of drug or dye will be used for this procedure.

SUMMARY:
In this study, study team aim to i) evaluate the accuracy of 3D IVS curvedness for prediction of RV systolic pressure (RVSP), mean pulmonary artery pressure (mPAP) and pulmonary vascular resistance (PVR) with RHC; ii) evaluate the usefulness of 3D IVS curvedness for predicting the response to vasodilator challenge with RHC, in patients clinically suspected or known to have primary PH.

DETAILED DESCRIPTION:
1) Pulmonary hypertension Pulmonary hypertension (PH) is manifested as an increase in mean pulmonary artery pressure (i.e., mPAP ≥ 25 mmHg) at rest on right heart catheterization (RHC) (Badesch 2009). It is a complex and multidisciplinary disorder causing restricted flow through the pulmonary arterial circulation due to increased pulmonary vascular resistance (PVR). It can be classified into five groups (Simonneau et al 2004): Group I - Idiopathic PAH, Familial PAH, and PAH associated with collagen vascular disease et al; Group II - PH with left heart disease; Group III - PH associated with lung diseases and/or hypoxemia; Group IV - PH due to chronic thrombotic and/or embolic disease; and Group V - miscellaneous causes of PH. The prognosis of PH is poor. The National Institutes of Health (NIH) Registry followed 194 patients with IPAH enrolled at 32 clinical centers from 1981 to 1985 (D'Alonzo et al 1991). The reported median survival rates of 68%, 48% and 34%. Similar results have been reported in Japan, India and Mexico.

Right heart catheterization (RHC) is the current reference standard for diagnosing PH (Galie et al 2009; McLaughlin et al 2009), according to ACCF/AHA expert consensus (McLaughlin et al 2009) and ESC/ERS guidelines (Galie et al 2009). Three hemodynamic measurements are essential from RHC: right ventricular systolic pressure (RVSP), mean pulmonary artery pressure (mPAP) and pulmonary vascular resistance (PVR). Further, patients with PH undergo RHC to assess clinical response to vasodilator challenge in order to guide therapy. It helps identify patients with better prognosis and patients who could potentially benefit from treatment with calcium channel blockers. A positive acute response is defined as a reduction of pulmonary artery pressure ≥10mmHg and ≤40mmHg. Although RHC plays a pivotal role in PH diagnosis, it is invasive and not without its own inherent risks (Hoeper et al 2006). For these reasons, development of a noninvasive alternative to RHC for diagnosis of PH is paramount.

Noninvasive diagnosis of PH and prediction of response to vasodilator challenge is clinically needed.

Several noninvasive methods for diagnosis of PH have been propounded, the most common being Doppler echocardiography. While routinely used to estimate pulmonary arterial pressure, Doppler measurement of tricuspid regurgitation jet peak velocity has inherent limitations: (i) the reliance on the visualization of the tricuspid regurgitant jet which is not always detectable, (ii) the fact that peak velocity of the jet may be difficult to measure in the presence of severe tricuspid regurgitation, and (iii) the need for adequate acoustic windows (Hinderliter et al 2003; Hachulla et al 2005). Furthermore, as recently emphasized in the ERS/ESC guideline (Galie et al 2009), estimation of mPAP or PVR must be an integral part of a complete cardiac echocardiographic examination.

It has long been recognized that systolic flattening and abnormal motion of the inter-ventricular septum (IVS), from either echocardiography (King et al 1983; Reisner et al 1994; Ricciardi et al 1999) or cine CMR images (Roeleveld et al 2005; Dellegrottaglie et al 2007; Alunni et al 2010), are signs of increased pulmonary arterial pressures. However, these studies are either qualitative or limited to 2D assessment, relying for analysis on subjective selection of the imaging plane and cardiac cycle phase. In the last 10 years, despite advances in biomedical engineering and computational approaches, no rigorous studies have been undertaken to study the relationship between quantitative 3D IVS shape and PH.

It is well documented that RV dysfunction and the 6-min walk test (6MWT) are associated with increased risk of mortality in PH (van Wolfersen 2007). Study team has recently developed a new method for assessment of RV function in terms of area strain, integrating radial, circumferential and longitudinal deformation (Zhong et al 2012). Therefore, we will also investigate the relationship between RV area strain and exercise capacity in PH.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to initiation of any study mandated procedure
* Age 16 years or more.
* Patient with clinically suspected or known primary PH belonging to one of the Updated Dana Point Clinical Classification Groups (I-IV)
* No known history of pulmonary hypertension

Exclusion Criteria:

Contraindication to MR examination:

* Cardiac pacemaker
* Brain aneurysm or clips
* Electronic implants or prosthesis
* Eye metal foreign body injury
* Severe claustrophobia

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 30 diagnosed pulmonary hypertension patient will be recruited from primary care clinic and outpatient clinics from the National Heart Centre Singapore.
  30 Healthy volunteer control.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-05; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
First occurrence of cardiovascular event. | 1-Year

CONTACTS AND LOCATIONS:
Overall Officials: Liang Zhong, PhD, Principal Investigator — National Heart Centre Singapore
Locations (1):
- National Heart Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leng S, Dong Y, Wu Y, Zhao X, Ruan W, Zhang G, Allen JC, Koh AS, Tan RS, Yip JW, Tan JL, Chen Y, Zhong L. Impaired Cardiovascular Magnetic Resonance-Derived Rapid Semiautomated Right Atrial Longitudinal Strain Is Associated With Decompensated Hemodynamics in Pulmonary Arterial Hypertension. Circ Cardiovasc Imaging. 2019 May;12(5):e008582. doi: 10.1161/CIRCIMAGING.118.008582. PMID 31088152